CLINICAL TRIAL: NCT00560651
Title: German Corneal Cross Linking Register
Status: Active, not recruiting | Type: Observational
Sponsor: Suphi Taneri (Other)
Responsible Party: Sponsor-Investigator, Suphi Taneri, Director, St. Franziskus Hospital
Organization: St. Franziskus Hospital (Other)
Other Study IDs: CCL
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Keratoconus
Keywords: keratoconus; cornea; cross linking; UV-light; riboflavin
MeSH Terms: conditions — Keratoconus; Corneal Diseases | interventions — Cefaclor; Corneal Cross-Linking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Cross linked eyes
  Interventions: Procedure: CCL (Corneal Cross Linking)

INTERVENTIONS:
Procedure: CCL (Corneal Cross Linking) — Apply Riboflavin 0.1% in Dextran 500 20% in NaCl solution Illuminate with UV-light of 365 nm wave-length and 3.0 mW/cm² intensity at 5 cm distance
  Other Names: Collagen cross linking; Corneal collagen cross linking; CCL; 3C-L

SUMMARY:
Corneal Cross Linking is new treatment modality for patients with keratoconus. A keratoconus is characterized by progressive bulging and thinning of the eye's cornea. Keratoconus is a potentially severely sight impairing condition that may necessitate corneal transplantation in the progressive state.

Corneal Cross Linking is designed to

* increase the cornea's mechanical stability
* to stop progression of bulging and thinning of the cornea
* to prevent the need for corneal transplantation

Corneal Cross Linking is performed by

1. Applying Riboflavin (Vitamin B2) eye drops every 2 minutes for 30 minutes to the cornea
2. Illuminating the cornea with UV-light

This register of Corneal Cross Linking procedures performed in Germany serves to

* gather long-term results
* detect rare complications and side-effects
* evaluate the efficacy in a large number of patients

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with keratokonus and treated with corneal cross Linking in Germany

Exclusion Criteria:

* Non-ectatic conditions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with Corneal Cross Linking in Germany
Sampling Method: Probability Sample
Enrollment: 7500 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2024-11 (Actual); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Keratometry | yearly

SECONDARY OUTCOMES:
Slit-lamp biomicroscopical findings | yearly
Best corrected Visual Acuity | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Suphi Taneri, MD, Study Chair — Augenklinik am St. Franziskus Hospital; Berthold Seitz, MD, Study Director — University of Homburg, Saar, Germany; Philip Maier, MD, Study Director — Univer. Freiburg, Germany; Claus Cursiefen, MD, Study Director — Univer. Erlangen, Germany; Thomas Reinhard, MD, Principal Investigator — Univers. Freiburg; Arnd Heiligenhaus, MD, Principal Investigator — Augenklinik am St.Franzsikus Hospital, Münster; Walter Sekundo, MD, Principal Investigator — Univers. Mainz; Theo Seiler, MD, Principal Investigator — IROC, Zürich; Atilla Osvald, MD, Principal Investigator — Univers Homurg, Saar; Jan M Vetter, MD, Principal Investigator — Univers. Mainz
Locations (2):
- Germany (2):
  - University of Saar, Homburg
  - Augenklinik am St. Franziskus Hospital, Münster

REFERENCES:
- [Background] Koller T, Seiler T. [Therapeutic cross-linking of the cornea using riboflavin/UVA]. Klin Monbl Augenheilkd. 2007 Sep;224(9):700-6. doi: 10.1055/s-2007-963492. German. PMID 17846959
- [Background] Spoerl E, Mrochen M, Sliney D, Trokel S, Seiler T. Safety of UVA-riboflavin cross-linking of the cornea. Cornea. 2007 May;26(4):385-9. doi: 10.1097/ICO.0b013e3180334f78. PMID 17457183
- [Background] Seiler T, Hafezi F. Corneal cross-linking-induced stromal demarcation line. Cornea. 2006 Oct;25(9):1057-9. doi: 10.1097/01.ico.0000225720.38748.58. PMID 17133053
- [Background] Wollensak G, Aurich H, Pham DT, Wirbelauer C. Hydration behavior of porcine cornea crosslinked with riboflavin and ultraviolet A. J Cataract Refract Surg. 2007 Mar;33(3):516-21. doi: 10.1016/j.jcrs.2006.11.015. PMID 17321404
- See also: Click here for more information about this study: German Register of Corneal Cross Linking — http://www.freiheit-ohne-brille.de